CLINICAL TRIAL: NCT04120181
Title: A New Predictor Marker for Cochlear Implants Infection: Neutrophil/ Lymphocyte Ratio
Brief Title: A New Predictor Marker for Cochlear Implants Infection
Status: Completed | Type: Observational
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Ozkan Onal, Professor, Selcuk University
Other Study IDs: 2019/01
Record Dates: First submitted 2019-10-07; First posted 2019-10-09 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Infection; Implant Infection; Cochlear Hearing Loss
Keywords: Neutrophil-to-lymphocyte ratio; Platelet-to-lymphocyte ratio; cochlear implant; artificial implant; infection
MeSH Terms: conditions — Infections; Hearing Loss, Sensorineural

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Control: The control group consists of 13 age- and gender-matched subjects who underwent CI surgery but showed no complications. The members of the control group were selected based on hospital records.
  Interventions: Other: There is no intervention.

INTERVENTIONS:
Other: There is no intervention. — There is no intervention.

SUMMARY:
Introduction: Surgical site infections associated with the cochlear implant can have serious consequences. Although advances in surgical techniques reduce these complications, it may be necessary to remove a device that works as a last resort as a result of ongoing infection. The removal of these devices, which are very expensive, increases the cost and takes the chance of hearing patients with this device. Therefore, it is very important to identify patients with a tendency to cochlear implant infection before surgery and to prevent these infections from occurring. Neutrophil/ lymphocyte ratio (NLR) and platelet/ lymphocyte ratio (PLR) are indicative of systemic inflammation and have a prognostic value in relation to mortality and morbidity in many diseases. The aim of this study was to identify patients with post-operative implant infection tendency in patients to be implanted with cochlear implant and to plan treatment for possible infections before cochlear implant, to reduce cost by preventing removal of implanted cochlear implant due to infection and to prevent the patient's chance of hearing through the cochlear implant from disappearing due to infection.

Methods: In this retrospective study, 13 patients with cochlear implant infection were included. Preoperative NLR was calculated by dividing the neutrophil (NEU) value by the lymphocyte (LYM) value and preoperative PLR was calculated by dividing the NEU value by the LYM value.

DETAILED DESCRIPTION:
A cochlear implant (CI) is a device that restores the sense of hearing in people with severe to profound hearing loss. This implant consists of two parts: The first is an internal component, which is surgically implanted under the skin behind the ear and connected to electrodes that are inserted inside the cochlea. The second is an external component that sits behind the ear and consists of a speech processor, a microphone, and a battery compartment. However, complications following device implantation may occur; these complications include flap erosion, local infections, general infections that may lead to meningitis, wound healing disorders, electrode insertion, device migration, and facial nerve injury (1,2). The incidence of infectious complications is quite uncommon, but potentially serious complication of CI surgery occurs at a rate of 1.7% to 4.1% (3-5). CI infection may be managed with conservative treatment modalities; however, persistent infection often ends in implant removal or implant replacement (6).

The body responds to inflammation and stress, including trauma, surgery, or sepsis, by elevating the neutrophil count and by reducing the lymphocyte count (7). Neutrophil/ lymphocyte ratio (NLR) is an indicator of poor prognostic factor in inflammation and in some diseases, such as obstructive sleep apnea syndrome, ischemic cardiac diseases, several types of cancer, and Bell's palsy (8-11). Platelet/ lymphocyte ratio (PLR) is also associated with inflammation and poor prognosis in patients with different types of cancer (12,13). Platelets release proinflammatory mediators, such as chemokines and cytokines (14). NLR and PLR can be calculated from complete blood count (CBC), a cheap and simple means of obtaining information regarding inflammation. During an inflammatory reaction, the amount of leukocytes in the circulation changes (9,15).

The relationship of preoperative NLR and PLR with CI infection has not yet been investigated and it is being aimed to show the predictive value of NLR and PLR in patients who developed implant infection after CI placement. First outcome is to compare whether there is a difference between NLR in patients with and without implant infection in patients with cochlear implant implantation. Secondary outcome is to determine which NLR is susceptible to infection if there is a difference between NLR between patients with and without implant infection.

ELIGIBILITY:
Inclusion Criteria:

1) Patients who developed implant infection after receiving cochlear implant at the Department of Otorhinolaryngology, Selcuk University Hospital between March 2014 - August 2018.

-

Exclusion Criteria:

1) Patients who had hematological disorders. 2) Diseases that retard tissue healing, such as diabetes, renal failure, or skin disease those who had experienced an impact on the head implant area.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study included 13 patients who developed implant infection after receiving cochlear implant at the Department of Otorhinolaryngology, Selcuk University Hospital between March 2014 - August 2018.
  The control group consists of 13 age- and gender-matched subjects who underwent CI surgery but showed no complications.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Difference between NLR in patients with and without implant infection | 2014-2018
  Our first outcome is to compare whether there is a difference between NLR in patients with and without implant infection in patients with cochlear implant implantation.

SECONDARY OUTCOMES:
Determine which NLR is susceptible to infection | 2014-2018
  Our Secondary outcome is to determine which NLR is susceptible to infection if there is a difference between NLR between patients with and without implant infection.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kanaan N, Winkel A, Stumpp N, Stiesch M, Lenarz T. Bacterial growth on cochlear implants as a potential origin of complications. Otol Neurotol. 2013 Apr;34(3):539-43. doi: 10.1097/MAO.0b013e3182829792. PMID 23478648
- [Background] Brady AJ, Farnan TB, Toner JG, Gilpin DF, Tunney MM. Treatment of a cochlear implant biofilm infection: a potential role for alternative antimicrobial agents. J Laryngol Otol. 2010 Jul;124(7):729-38. doi: 10.1017/S0022215110000319. Epub 2010 Mar 10. PMID 20214837
- [Background] Wei BP, Shepherd RK, Robins-Browne RM, Clark GM, O'Leary SJ. Threshold shift: effects of cochlear implantation on the risk of pneumococcal meningitis. Otolaryngol Head Neck Surg. 2007 Apr;136(4):589-96. doi: 10.1016/j.otohns.2006.11.039. PMID 17418257
- [Background] Zahorec R. Ratio of neutrophil to lymphocyte counts--rapid and simple parameter of systemic inflammation and stress in critically ill. Bratisl Lek Listy. 2001;102(1):5-14. English, Slovak. PMID 11723675
- [Background] Seretis C, Gourgiotis S, Gemenetzis G, Seretis F, Lagoudianakis E, Dimitrakopoulos G. The significance of neutrophil/lymphocyte ratio as a possible marker of underlying papillary microcarcinomas in thyroidal goiters: a pilot study. Am J Surg. 2013 Jun;205(6):691-6. doi: 10.1016/j.amjsurg.2012.08.006. Epub 2013 Feb 4. PMID 23388425
- [Background] Senturk M, Azgin I, Ovet G, Alatas N, Agirgol B, Yilmaz E. The role of the mean platelet volume and neutrophil-to-lymphocyte ratio in peritonsillar abscesses. Braz J Otorhinolaryngol. 2016 Nov-Dec;82(6):662-667. doi: 10.1016/j.bjorl.2015.11.018. Epub 2016 Mar 28. PMID 27068888
- [Derived] Onal M, Colpan Keles B, Ulusoy B, Onal O. New validation of a well-known marker in cochlear implant infections: A retrospective, case-controlled, observational study. Laryngoscope Investig Otolaryngol. 2022 Nov 24;7(6):1992-2001. doi: 10.1002/lio2.900. eCollection 2022 Dec. PMID 36544965